CLINICAL TRIAL: NCT00325286
Title: Open Label Prophylaxis Study of Lithium Plus Extended- Release Carbamazepine (Equetro®) Combination for Rapid Cycling Bipolar Disorder
Brief Title: Open Label Study of Lithium Plus Extended-Release Carbamazepine (ERC-CBZ) for Rapid Cycling Bipolar Disorder
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Creighton University (Other)
Collaborators: Shire (Industry)
Responsible Party: Sriram Ramaswamy, M.D., Assistant Professor of Psychiatry, Creighton University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-13934
Record Dates: First submitted 2006-05-10; First posted 2006-05-12 (Estimated); Last update posted 2007-12-14 (Estimated); Status verified 2007-12

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Lithium; Carbamazepine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Treatment with lithium and extended release carbamazepine
  Interventions: Drug: Lithium Plus Extended- Release Carbamazepine

INTERVENTIONS:
Drug: Lithium Plus Extended- Release Carbamazepine — Preliminary phase subjects receive ERC-CBZ starting dose range from 100 to 200 mg b.i.d. and further titration up to a maximum dose of 1600 mg/day done at the discretion of the investigator. Titration phase will not extend beyond 2 weeks.Open label phase subjects stabilized on lithium and ERC-CBZ therapy will enter this phase for 6 months
  Other Names: Epitol, Tegretol

SUMMARY:
This is an open label design using Lithium plus extended release carbamazepine (Equetro) in combination for 6 months. Rapid cycling bipolar disorder is frequently treatment refractory and associated with repeated hospitalizations and complications. The results of this study will offer a promising approach to treat this complex disorder. The primary efficacy measure will be the time to relapse. Relapse will determined by the investigator based on the following: Need for additional pharmacotherapy for mood-related symptoms, hospitalization for an mood episode, increase of more than 50% in HAM-D and YMRS scores from the baseline visit.

DETAILED DESCRIPTION:
Open label Design with Lithium plus Extended release carbamazepine combination for 6 months. Extended release carbamazepine at doses of 1600 mg/day will be utilized. Lithium dosage will be adjusted to maintain therapeutic blood levels.

Patient Population: N = 20.

Primary and Secondary Efficacy Endpoints:

The primary efficacy measure will be the time to relapse. Relapse will determined by the investigator based on the following

* Need for additional pharmacotherapy for affective symptoms
* Hospitalization for an affective episode
* Increase of more than 50% in HAM-D and YMRS scores from baseline

The differences in the frequency of affective episodes in the 6-month prior to the treatment with ERC-CBZ and 6 months after treatment initiation will also be measured. Secondary efficacy measures will include; changes in the 17- Item Hamilton Depression Scale (HAM-D), Young Mania Rating Scale (YMRS), Clinical Global Severity Scale (CGI -S), Clinical Global Improvement Scale (CGI-I) scores at baseline and scores during treatment with ERC-CBZ.

Inclusion Criteria:

1. Subjects, 19 years and older with DSM-IV defined Bipolar Disorder with a history of the rapid cycling within the past 12 months.
2. Subjects may be either in a manic, mixed or depressive phase at time of study entry.
3. Subjects must be on lithium therapy for 6 months or longer. Stable lithium therapy will be defined as: No changes in lithium dosage for at least 2 weeks prior to study entry and a therapeutic lithium level (0.6 to 1.2 mEq) prior to study entry.

Exclusion Criteria:

1. Subjects with a lifetime history of Schizophrenia or Schizoaffective Disorder
2. If patients are on thyroid replacement therapy they have to on stable doses for the past 3 months at study enrollment.
3. Presence of active suicide ideations or score of > 3 on the suicide subscale of the 17 - item HAM-D.
4. Current substance dependence (excluding nicotine) defined as no dependence criteria for 30 days prior to study enrollment
5. Subjects with a history of non-response to carbamazepine or lithium
6. Subjects who are pregnant or planning to become pregnant
7. Subjects with a history of allergic/idiosyncratic reaction or intolerability to carbamazepine or lithium.

Study Procedures:

Preliminary Phase: The Structured Clinical Interview Diagnostic Schedule (SCID), medical & psychiatric history and baseline laboratory testing, EKG; pregnancy test will be obtained to ensure study eligibility. Eligible subjects will receive ERC-CBZ at starting doses ranging from 100 to 200 mg b.i.d. depending on clinical presentation and further titration up to a maximum dose of 1600 mg/day will be done at the discretion of the investigator. This titration phase will not extend beyond 2 weeks during which changes in concomitant medications will be allowed. Next, all psychotropics excluding lithium, ERC-CBZ and benzodiazepines will be tapered over a 2-week period. During the preliminary phase subjects will be seen weekly and assessments will be made using the HAM-D, YMRS, CGI -S, CGI-I, AE, and Concomitant medications

Open Label Phase: Subjects on lithium and ERC-CBZ therapy will enter this phase for 6 months. Changes to both lithium and ERC-CBZ will be permitted during this phase with serum levels to guide titration. Use of lorazepam, as a rescue medication will be permitted. Study visits will be every biweekly for 6 months. The HAM-D, YMRS and CGI-S, CGI-I, AE, concomitant medications will be assessed at each visit. Compliance will be assessed by pill counts at each study visit.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects, 19 years and older with DSM-IV defined Bipolar Disorder with a history of the rapid cycling within the past 12 months.
2. Subjects may be either in a manic, mixed or depressive phase at time of study entry.
3. Subjects must be on lithium therapy for 6 months or longer. Stable lithium therapy will be defined as: No changes in lithium dosage for at least 2 weeks prior to study entry and a therapeutic lithium level (0.6 to 1.2 mEq) prior to study entry.

Exclusion Criteria:

1. Subjects with a lifetime history of Schizophrenia or Schizoaffective Disorder
2. If patients are on thyroid replacement therapy they have to on stable doses for the past 3 months at study enrollment.
3. Presence of active suicide ideations or score of > 3 on the suicide subscale of the 17 - item HAM-D.
4. Current substance dependence (excluding nicotine) defined as no dependence criteria for 30 days prior to study enrollment
5. Subjects with a history of non-response to carbamazepine or lithium
6. Subjects who are pregnant or planning to become pregnant
7. Subjects with a history of allergic/idiosyncratic reaction or intolerability to carbamazepine or lithium.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-05; Study Completion 2008-03 (Estimated)

PRIMARY OUTCOMES:
The primary efficacy measure will be the time to relapse. Relapse will determined by; need for additional pharmacotherapy, hospitalization for an affective episode, increase of >/= 50% in HAM-D and YMRS scores. | Patients will be seen weekly during preliminary phase and biweekly during the open label phase

SECONDARY OUTCOMES:
The differences in the frequency of affective episodes in the 6-month prior to the treatment with ERC-CBZ and 6 months after treatment initiation will also be measured. Secondary efficacy measures will include; changes in the 17- Item Hamilton Depression | Patients will be seen weekly during the preliminary phase and biweekly during the open label phase

CONTACTS AND LOCATIONS:
Overall Officials: Sriram Ramaswamy, M.D., Principal Investigator — Creighton University
Locations (1):
- Creighton University Department of Psychiatry, Omaha, Nebraska, United States